CLINICAL TRIAL: NCT05351151
Title: Analgesic Efficacy of Echoguided Maxillary and Mandibular Nerve Blocks in Planned Maxillomandibular Osteotomy Surgery
Brief Title: Pain Reduction in Maxillomandibular Surgery Using Maxillary and Mandibular Nerve Blocks
Acronym: ECHOMAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/21/0509
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-02

CONDITIONS: Pain, Post Operative; Regional Anesthesia
Keywords: Orthognathic surgery; Maxillary-mandibular osteotomy; Double jaw osteotomy; Bimaxillary surgery; Maxillary nerve block; Mandibular nerve block; Regional anesthesia; Nerve blocks
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loco Regional anesthesia (LRA) (Experimental): The LRA group is made up of patients benefiting from the V2 and V3 ultrasound-guided LRA technique without mucosal infiltration.
  Interventions: Procedure: bilateral ultra-sound guided maxillary and mandibular nerve blocks
- Infiltration (Active Comparator): The "Infiltration" group is made up of patients who benefit from the infiltration technique by local anesthesia of the incision sites by the surgeon without recourse to ultrasound-guided LRA.
  Interventions: Procedure: Infiltration of Lidocaine 1%

INTERVENTIONS:
Procedure: bilateral ultra-sound guided maxillary and mandibular nerve blocks — Interventional group will receive bilateral ultra-sound guided maxillary and mandibular nerve block with ROPIVACAINE 4,75 mg/ml.
  Arms: Loco Regional anesthesia (LRA)
Procedure: Infiltration of Lidocaine 1% — Intervention requiring the infiltration of LIDOCAINE 1% at incision sites by surgeon after general anesthesia induction during maxillo-mandibular osteotomy
  Arms: Infiltration

SUMMARY:
Maxillo-mandibular osteotomy is a painful surgery which requires mostly opioids use. Recent studies on maxillary and mandibular nerve blocks have suggested benefit in maxillo-facial surgery but have been poorly investigated in orthognathic surgery. This study is designed to evaluate analgesic effectiveness, through opioids consumption, of a bilateral double ultra-sound guided nerve blocks (maxillar and mandibular nerve) in maxillo-mandibular osteotomy.

DETAILED DESCRIPTION:
Maxillo-mandibular osteotomy is a frequent but painful procedure in maxillo-facial surgery. It mostly requires opioids use which lead to well known side effects. Regional anesthesia has strongly modified post-surgical rehabilitation of many procedures. Maxillary nerve block has proved its efficiency on opioid consumption reduction in pediatric cleft palet surgery but has been rarely evaluated in orthognathic surgery. Mandibular nerve block has never been investigated in maxillo-mandibular osteotomy as well as benefit of bilateral ultra-sound guided technique to perform these nerve blocks. Consequently, this trial is designed to evaluate analgesic effectiveness of a double ultra-sound guided nerve blocks (maxillar and mandibular nerve) in maxillo-mandibular osteotomy.

This monocentric, single-blinded, randomized controled trial is designed with 2 groups of 25 patients receiving either bilateral double ultra-sound guided nerve block (maxillary and mandibular) with ROPIVACAINE 4.75mg/mL either local infiltration of LIDOCAINE 1% at incision sites by surgeon after general anesthesia induction during maxillo-mandibular osteotomy. Per et post-surgery anesthesic protocol and analgesia are standardized for both group. The main outcome corresponds to opioid consumption in MME of the first 24h after surgery. Follow-up occurs at 24h and 48h after end of surgery to assess analgesia, pain and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 15 to 45 years old,
* Scheduled for maxillary-mandibular osteotomy,
* Registered in French social insurance register,
* With informed consent disclosure.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification ≥ 3
* Innate or acquired hemostasis pathology,
* Peripheric neuropathy,
* Drug intake for chronic pain,
* Infection/scar at needle insertion site,
* Associated rhinoplasty surgery,
* Allergy to local anesthetics,
* Pregnant woman or potentially,
* Breastfeeding woman,
* Already registered in other clinical trial,
* Adults under legal protection of incapable adult,
* Cognitive disease impairing using of evaluation tools performed in protocol,
* All contraindication of anesthetics drugs used in protocol.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
The opioid consumption (in Morphine Milligram Equivalents) after the first 24 hours post-surgery. | 24 hours post-surgery
  The opioid consumption (in Morphine Milligram Equivalents ) after the first 24hours post-surgery.

SECONDARY OUTCOMES:
Opioid consumption in Morphine Milligram Equivalents after the first 48 hours post-surgery. | 48 hours post-surgery
  Evaluation of the total consumption of morphine equivalents (Oxycodone Hydrochloride) after the first 48 hours postoperative hour.
Maximal pain (Numerical Rating Scale) in recovery room, at 24h after surgery. | 24 hours after surgery
  Pain assessment by Simple Numerical Scale (ENS from 0 to 10) in the Postoperative Monitoring Room (maximum value) at the 24th postoperative hour
Maximal pain (Numerical Rating Scale) in recovery room, at 48 hours after surgery. | 48 hours after surgery
  Pain assessment by Simple Numerical Scale (ENS from 0 to 10) in the Postoperative Monitoring Room (maximum value) at the 48th postoperative hour.
Incidence of opioid-Emergent Adverse Events [Safety and Tolerability] | 3 days
  Measuring the incidence rate of common side effects associated with morphine drugs
Evaluation of preoperative anxiety and fear using Amsterdam Preoperative Anxiety and Information Scale on post-surgical pain | pré-anesthesic visit (day -1 or day 0)
  The patient's degree of pre-operative anxiety will be assessed using the Amsterdam Preoperative Anxiety and Information questionnaire in French Items are rated on a 5-point Likert scale ranging from 1 = "not at all" to 5 = "extremely"
Evaluation of patient satisfaction about medical care | 3 days (maximum)
  The patient's feelings and satisfaction with their care will be evaluated by completing the questionnaire The feeling and satisfaction is rated according to a scale of 5 categories as follows: None, Low, Medium, High and Very High
Incidence of regional anesthesia-Emergent Adverse Event [Safety and Tolerability] | 3 days
  Measuring the incidence rate of common side effects associated with regional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marion MURE, Ph, Principal Investigator — University hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

REFERENCES:
- [Result] Esquerre T, Mure M, Minville V, Prevost A, Lauwers F, Ferre F. Bilateral ultrasound-guided maxillary and mandibular combined nerves block reduces morphine consumption after double-jaw orthognathic surgery: a randomized controlled trial. Reg Anesth Pain Med. 2025 Jul 4;50(7):575-580. doi: 10.1136/rapm-2024-105497. PMID 38697776